CLINICAL TRIAL: NCT06101004
Title: A Multi-center, Non-interventional Prospective Clinical Trial to Evaluate the Safety and Effectiveness of CVA-FLOW Software Device for the Detection of Stroke and LVO in Patients With Suspected Stroke
Brief Title: A Multi-center, Non-interventional Prospective Clinical Trial to Evaluate the Safety and Effectiveness of CVA-FLOW
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cvaid Medical (Industry)
Collaborators: Donawa Lifescience Consulting (Unknown)
Responsible Party: Sponsor
Other Study IDs: CVA-001
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: emergency department; LVO
MeSH Terms: conditions — Stroke; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CVA-Flow — CVA-FLOW Software Device is indicated for the detection of Stroke and LVO in patients with suspected stroke.

SUMMARY:
CVAid Medical Ltd. developed a smartphone-based tele stroke system named CVA-Flow. This system aims to evaluate the patient's neurological status, particularly detection of a possible stroke, assessment of stroke severity, and prediction of LVO as the cause of stroke. The system's app guides the user through the examination step by step based on NIHSS/ Rapid Arterial Occlusion Evaluation (RACE) scales. The video can also be transferred offline to enable a distant stroke physician to assess the patient's status manually.

DETAILED DESCRIPTION:
Management of acute ischemic stroke has changed dramatically following the evidence of the superiority of endovascular treatment (EVT) over best medical management, in the treatment of patients suffering large vessel occlusion (LVO), within 24 hours from onset of symptoms. The immediate consequence was an increase in the number of patients eligible for EVT, requiring secondary transfer of those patients from primary stroke centers to comprehensive stroke centers, capable of performing EVT.

EVT requires accurate and rapid diagnosis in the prehospital setting, as it is only indicated in specific patients with LVO, making up a small percentage of stroke cases, and its beneficial effects are highly time-dependent.

Of the existing diagnostic tools that accurately distinguish LVO cases from non-LVO ones, the National Institutes of Health Stroke Scale (NIHSS) is the most recommended tool by healthcare providers to objectively quantify the neurological impairment caused by a suspected stroke. Nevertheless, the NIHSS is not considered to be feasible in the pre-hospital setting of EMS, since it requires a greater degree of training, is thought to be too time-consuming, and has not been as well validated in the prehospital setting.

Several previous studies showed feasibility and reliability of the use of telemedicine for determining the NIHSS score from afar in stroke patients in real time, in simulated stroke patients in real time and captured video segments. Previous studies did not use designated applications designed for performing neurological evaluations, relying on simple applications for video conferencing instead, therefore requiring applicators to possess knowledge in performing neurological examinations and evaluators to be online the whole examination time.

To resolve this issue, CVAid Medical Ltd. developed a smartphone-based tele stroke system named CVA-Flow. This system aims to evaluate the patient's neurological status, particularly detection of a possible stroke, assessment of stroke severity, and prediction of LVO as the cause of stroke. The system's app guides the user through the examination step by step based on NIHSS/ Rapid Arterial Occlusion Evaluation (RACE) scales. The video can also be transferred offline to enable a distant stroke physician to assess the patient's status manually.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years of age
* With suspected acute stroke at the ED prior to treatment (tPA or EVT)

Exclusion Criteria:

* Patient intubated upon arrival
* Patient treated with tPA prior to arrival at the ED
* Patients with the following conditions:

  * Brain tumors
  * Hypoglycemia
  * Toxic poisoning
  * Seizures
  * Sepsis
  * Subdural hematoma
  * Encephalopathy (uremic, hepatic or other)
  * Encephalitis
* Previous stroke with permanent neurological deficit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected acute stroke at the ED prior to treatment (tPA or EVT)
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Co-primary endpoints are defined to demonstrate the performance of CVA-Flow to detect patients with stroke among all suspected patients. | From the time of recruitment of the subject to discharge from hospital estimated to be up to 4 weeks
  The co-primary endpoints are defined as follows,
  Reference for each case shall be scored by the reviewer neurologist dichotomously as:
  * Positive - at least one relevant finding, or;
  * Negative - no relevant findings.
  Each case shall also be scored dichotomously by CVA-Flow software as:
  * Positive - suspected stroke, or;
  * Negative - no suspected stroke.

SECONDARY OUTCOMES:
Confirmatory secondary endpoints are defined to demonstrate the performance of CVA-Flow to detect patients with LVO stroke among all suspected patients without head bleeding. | From the time of recruitment of the subject to discharge from hospital estimated to be up to 4 weeks
  The confirmatory secondary endpoints are defined similarly to the co-primary endpoints as follows,
  Reference for each case shall be scored by the reviewer radiologist dichotomously as:
  * Positive - at least one relevant finding (LVO), or;
  * Negative - no relevant findings.
  Each case shall also be scored dichotomously by CVA-Flow software as:
  * Positive - suspected LVO, or;
  * Negative - no suspected relevant findings.

CONTACTS AND LOCATIONS:
Locations (2):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Hospital Vall d'Hebron - Neurology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No